CLINICAL TRIAL: NCT02717468
Title: Comparative Noninvasive Continuous Cardiac Output by the Clearsight With Invasive Monitoring by Pulsioflex in Abdominal Surgery
Acronym: CLEARSIGHT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2015-A01895-44
Record Dates: First submitted 2016-02-18; First posted 2016-03-23 (Estimated); Last update posted 2018-05-18 (Actual); Status verified 2016-10

CONDITIONS: Cardiac Output Measurement
MeSH Terms: interventions — Cardiac Output

INTERVENTIONS:
Device: Cardiac output and stroke ejection volume monitoring with arterial waveform analysis in the digital artery (ClearSight®)
Device: Cardiac output and stroke ejection volume monitoring with arterial waveform analysis in the radial artery (Pulsioflex®).

SUMMARY:
In high-risk patients, it is now recommended to guide the intraoperative volume replacement via the stroke volume.

Today, the most commonly used technique for estimating the stroke volume is the arterial waveform analysis in the radial artery. This technique has the disadvantage of being invasive and increasing the time dedicated to anesthesia during the surgery.

The future is the non-invasive monitoring of stroke volume. Thus, Edwards Life Science has developed a continuous monitoring technology and non-invasive arterial pressure, cardiac output and stroke volume using a digital sensor (ClearSight®). The continuous monitoring of blood pressure by this technique was validated in cardiothoracic surgery but studies about monitoring cardiac output or stroke volume are inconclusive and contradictory.

The objective of this study is to compare the use of non-invasive monitoring of stroke volume by Clearsight® with the arterial waveform analysis in the radial artery by Pulsioflex® in major surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo major surgery
* Patients monitored by a Pulsioflex® device

Exclusion Criteria:

* Patients with heart rhythm disorder
* Patients with Raynaud's disease or vasculitis
* Emergency surgery
* Significant edema fingers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-02; Primary Completion 2016-12 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Stroke Ejection Volume (SEV) measure by ClearSight® | 24 hours
Stroke Ejection Volume (SEV) measure by Pulsioflex® | 24 hours

SECONDARY OUTCOMES:
Cardiac Output (CO) measure by ClearSight® | 24 hours
Cardiac Output (CO) measure by Pulsioflex® | 24 hours
Stroke Ejection Volume Variations (SVV) measure by ClearSight® | 24 hours
Stroke Ejection Volume Variations (SVV) measure by Pulsioflex® | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Matthieu BOISSON, Poitiers, France